CLINICAL TRIAL: NCT02558699
Title: Clinical Usefulness of Virtual Ablation Guided Catheter Ablation of Atrial Fibrillation: Virtual Rotor Mapping and Catheter Ablation
Acronym: CUVIA-AF II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2015-0646
Record Dates: First submitted 2015-09-23; First posted 2015-09-24 (Estimated); Last update posted 2023-01-03 (Actual); Status verified 2022-12

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional group (Active Comparator): Group operating the atrial fibrillation by physician's personal experience, not by virtual simulation.
  Interventions: Procedure: physician's personal experience
- 3D atrial computer model (Experimental): Group choosing choose the best effective rotor mapping by simulating 3D atrial computer model which consider patinet's heart size and shape.
  Interventions: Procedure: Virtual rotor mapping

INTERVENTIONS:
Procedure: physician's personal experience — physician's personal experience
  Arms: conventional group
Procedure: Virtual rotor mapping — Virtual rotor mapping
  Arms: 3D atrial computer model

SUMMARY:
Radiofrequency catheter ablation is effective in the treatment of patients with paroxysmal atrial fibrillation. In order to reduce the recurrence rate after catheter ablation, the investigators propose to apply 'virtual' ablation on patient-specific atria by simulating 3D atrial computer model. The investigators will conduct virtual rotor mapping in the patient specific atrial model. Then, the investigators will compare the clinical outcome of conventional circumferential pulmonary vein isolation and additional rotor ablation guided by virtual rotor mapping.

ELIGIBILITY:
Inclusion Criteria:

* AF patient age 19~80
* Diagnosis of AF patients who performed catheter ablation of atrial fibrillation due to uncontrolled pulse rate by anti-arrhythmic drug therapy.

Exclusion Criteria:

* AF patients who have severe heart deformations or vascular disease.
* The patient who have renal disease of eGFR<30mL/min
* The patients who had been performed catheter ablation of atrial ablation and MAZE.
* The patients who missed out to recording of 3D CT, echo and electrocardiography.
* the patient have experienced major hemorrhagic complication
* The patient have experienced ischemic cerebral infarction more 2 times
* The patient who have risk of ischemic cerebral infarction (CHA2DS2-VASc Score >5)

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2018-08-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of atrial fibrillation of 18 months after procedure within 18 months | 18 months
Rate of mortality, incidence of cerebral infarction and hospitalization after procedure | 24 months

SECONDARY OUTCOMES:
Major complication related procedure : Complication of hemorrhagic and embolic | 24 months
Pericardial effusion required treatment, 4g/dL reduced level of Hb, Hemorrhage required blood transfusion and Cerebral infarction related procedure | 24 months
Procedure time and Radiofrequency ablation time | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University Health System, Seoul, South Korea

REFERENCES:
- [Derived] Choi Y, Lim B, Yang SY, Yang SH, Kwon OS, Kim D, Kim YG, Park JW, Yu HT, Kim TH, Yang PS, Uhm JS, Shim J, Kim SH, Sung JH, Choi JI, Joung B, Lee MH, Kim YH, Oh YS, Pak HN; CUVIA-REGAB Investigators. Clinical Usefulness of Virtual Ablation Guided Catheter Ablation of Atrial Fibrillation Targeting Restitution Parameter-Guided Catheter Ablation: CUVIA-REGAB Prospective Randomized Study. Korean Circ J. 2022 Sep;52(9):699-711. doi: 10.4070/kcj.2022.0113. Epub 2022 Jul 11. PMID 35927040